CLINICAL TRIAL: NCT00279513
Title: A Randomised, Double- Blind, Placebo Controlled, Clinical Trial to Assess the Efficacy of the Homeopathic Medication TRAUMEEL S in Reducing Pain After Surgical Correction of Hallux Valgus
Brief Title: TRAUMEEL S in Reducing Pain After Correction of Hallux Valgus-Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Menachem Oberbaum, MD, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HV-2006
Record Dates: First submitted 2006-01-09; First posted 2006-01-19 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-04

CONDITIONS: Post Hallux Valgus Repair Pain
Keywords: homeopathy; hallux valgus; pain; traumeel s
MeSH Terms: conditions — Hallux Valgus; Pain | interventions — Traumeel S

INTERVENTIONS:
Drug: Traumeel S

SUMMARY:
Hallux valgus is a common deformity of the big toe, defined as medial deflection of the first metatarsal bone along with lateral deflection of the first toe. Surgery has been shown to be beneficial when compared to orthoses or no treatment. While generally effective, surgery entails significant post-operative pain, inflammation and edema, and several weeks of limited mobility. This will be a double-blind, randomized, placebo-controlled study comparing the homeopathic drug Traumeel S with placebo in pain reduction after surgical Hallux valgus correction.

80 patients, over the age of 18 years, undergoing surgical correction of unilateral hallux valgus will be enrolled in the trial. The patients will be randomized to two groups, one receiving oral Traumeel S and the other oral placebo tablets. Patients will take active or placebo medication for 13 days or until they have a NRS score of 3 or less for 2 consecutive days. Pain will be reported daily by the patient on the patient diary, using an 11-point numerical rating score (NRS-11) during 13 days post-operatively. They will also be asked to report daily consumption of primary and "rescue" analgesics for 13 days post-operatively. Patients will be contacted daily by the research assistant to encourage compliance and to record their daily NRS and analgesic consumption in the CRF. Patients will be evaluated by physicians at six and 13 days postoperatively for redness and compliance.

ELIGIBILITY:
Inclusion Criteria:

Patients of either sex undergoing unilateral surgical correction of Hallux Valgus.

Age over 18 years. Signature upon informed consent form. Meeting none of exclusion criteria.

Exclusion criteria Participation in another clinical trial within 4 weeks prior to enrollment. Inability to comply with the study protocol. Previous surgical Hallux Valgus correction on ipsilateral foot. Current use of analgesia for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Pain

SECONDARY OUTCOMES:
Analgesics consumed
Days of "rescue" analgesic use
Area of redness
The safety treatment

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Oberbaum, M.D., Principal Investigator — Shaare Zedek Medical Center, Jerusalem, Israel
Locations (1):
- Dept. of Orthopedic Surgery, Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Derived] Singer SR, Amit-Kohn M, Weiss S, Rosenblum J, Maoz G, Samuels N, Lukasiewicz E, Freedman L, Paltiel O, Itzchaki M, Niska M, Oberbaum M. Traumeel S for pain relief following hallux valgus surgery: a randomized controlled trial. BMC Clin Pharmacol. 2010 Apr 12;10:9. doi: 10.1186/1472-6904-10-9. PMID 20380750